CLINICAL TRIAL: NCT06603727
Title: Combined Cognitive and Physical Training for the Neurorehabilitation of Patients With Cognitive Deficits Due to the Human Immunodeficiency Virus: a Pilot Study
Brief Title: Computerized Cognitive Rehabilitation of Patients With Cognitive Deficits Due to the Human Immunodeficiency Virus
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Principal Investigator, Prof. Arseny Sokolov, MD, PhD, Professor, MD, Centre Hospitalier Universitaire Vaudois
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CHUV-DNC-CCT-HIV-2022
Record Dates: First submitted 2024-08-12; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Human Immunodeficiency Virus; Cognitive Dysfunction
Keywords: HIV Infections; Communicable Diseases; Neurological Rehabilitation; Cognitive Behavioural Therapy; Exercise Therapy; Nervous System Diseases; Neurocognitive Disorders; Cognition Disorders; Mental Disorders
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Cognitive Dysfunction; HIV Infections; Communicable Diseases; Nervous System Diseases; Neurocognitive Disorders; Cognition Disorders; Mental Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Masking will affect participants and study personnel, with exception to the personnel supervising the training programs.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Program 1 (Experimental): Computerized Gaming Rehabilitation Program 1
  Interventions: Device: Computerized Gaming Rehabilitation Program 1
- Program 2 (Active Comparator): Computerized Gaming Rehabilitation Program 2
  Interventions: Device: Computerized Gaming Rehabilitation Program 2

INTERVENTIONS:
Device: Computerized Gaming Rehabilitation Program 1 — Brain training games displayed on a large screen paired with physical exercise component. The program involves movements such as reaching, stepping, or stretching in place.
  Arms: Program 1
Device: Computerized Gaming Rehabilitation Program 2 — Brain training games displayed on a tablet device paired with physical exercise component. The program involves movements such as reaching, stepping, or stretching.
  Arms: Program 2

SUMMARY:
WHO: 24 participants with cognitive deficits due to a Human Immunodeficiency Virus (HIV) infection, able to engage in moderate physical activity.

WHY: The Human Immunodeficiency Virus is known to cause deficits in cognitive function, even under effective pharmacological viral load suppression. Cognitive dysfunction in patients with HIV is frequent and has a detrimental impact on their everyday personal and professional life. The purpose of this study is to evaluate two sets of computerized exercises combining cognitive and physical effort to see if they can improve executive function in patients with an HIV infection.

WHAT: Study participants first undergo cognitive and physical assessments. Additional questionnaires will assess mood, everyday life cognition, function and quality. This will be followed by a 6 week training period with 2 training sessions a week. The effect of the physical and cognitive training will be measured in a post-training evaluation session. Six months after completion of the training, the study will evaluate cognitive and physical abilities of participants to study long-term effects of the respective training program.

WHERE: Both the evaluation and the training sessions will be conducted on the premises of the Lausanne University Hospital (Rue du Bugnon 46, 1005 Lausanne, Switzerland)

DETAILED DESCRIPTION:
This is an exploratory Randomized Controlled Trial with the purpose of evaluating the potential of two sets of gamified cognitive and physical exercises in the neurorehabilitation of cognitive deficits due to an infection with the Human Immunodeficiency Virus (HIV).

Upon recruitment, eligible study participants (see 'Eligibility Criteria') receive a detailed oral and written description about the scientific background, aims and methods of the study. Additional information will be provided about potential benefits and risks associated with study participation, as well as about the voluntary nature of participation throughout the study. The participant's written informed consent is required for study enrollment.

After inclusion in the study, participants are randomized into one of two different training programs with equal chance of attribution and without possibility of choosing:

* Program 1 involves brain training and guided, light physical exercise games on a tablet device. The exercise involves movements such as reaching, stepping, and stretching. Warm-up and cool down sessions are mandated prior to and following the tasks.
* Program 2 involves gamified exercises displayed on a large screen. Participants use whole-body movements to complete the tasks. Tasks involve movements such as reaching, stepping, and jogging in place. These movements are tracked by a motion sensor. Warm-up and cool down sessions are mandated prior to and following the training sessions.

Independently of program attribution, participants engage in a pre-training assessment, a six-week training period, a post-training assessment and a 6-month-follow-up assessment.

Before the start of the training, participants are required to perform several cognitive and physical tests (including cyclo-ergospirometry) and fill out a number of questionnaires on subjective cognitive function, mood and quality of life. Additionally, an electroencephalography (EEG) will be performed to measure brain activity. The exercises, the questionnaires and the EEG serve as a baseline evaluation of cognitive, physical and neurophysiological function.

Following the first assessment, study participants engage in a six-week training period. In both programs, participants engage in two weekly trainings of ninety minutes duration each.

After completion of the training period, study participants engage in a post-training assessment to evaluate the effect of training on cognitive and physical performance. This session incorporates the same tasks and questionnaires as in the pre-training visit. An EEG will be used to characterize the training effects on dynamics of the underlying large-scale neuronal networks. The aim of the post-training assessment is to demonstrate immediate training effect of the two programs.

A final follow-up visit is scheduled 6 months after the completion of the last training session. The cognitive and physical testing together with the questionnaires and the EEG will be repeated to examine the long-term effects of the training programs.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Diagnosis of an HIV infection
* Undetectable HIV load in the serum (<50 copies/mL) over the last 6 months prior to study inclusion.
* Z-score ≤ -1.0 in at least one of the three following tests:

  * Color Trail Test (CTT) Flexibility Index
  * subtest Code of the Wechsler Adult Intelligence Scale - Fourth Edition (WAIS-IV)
  * subtest Digit Span of the WAIS-IV
* Z-score ≤ -1.0 in at least one of the following tests:

  * Symbol Digits Modalities Test (SDMT)
  * Brief Visuospatial Memory Test Revised (BVMT-R)
  * CTT Flexibility Index
  * Stroop Color-Word interference test

Exclusion Criteria:

* Clinically defined cause for cognitive deficits other than HIV
* Diagnosis of severe depression according to a cut-off score of ≥ 27 of the Center for epidemiological studies - depression questionnaire (CES-D; Metral et al., 2020; Radloff, 1977)
* Diagnosis of HIV-associated dementia according to the Frascati Critera (Antinori et al., 2007)
* Current psychotic symptoms according to the Mini-International Neuropsychiatric Interview (M.I.N.I. - L, Sheehan et al., 1998) subscale of psychotic symptoms
* Antidepressive, anxiolytic or cART medication that has been changed over the last month
* Thoracic pain and/or heart palpitations at rest, during or following a physical effort (based on self-report)
* For patients without known and clinically stable cardio-vascular disease: abnormal rest electrocardiogram readings suggestive of second degree type Mobitz or third degree atrioventricular blocking, pathological repolarization (T-wave inversion, ST elevation, abnormal QT lengthening in at least two corresponding leads), or typical features of channelopathies
* Premature termination of maximal effort test due to cardiac problems
* Falls in the past 12 weeks as evaluated in the enrolment interview (Hopkins Falls Grading Scale, Grade >1)
* High risk of falling according a cutoff score > 15 sec in the Four Square Step Test (Dite & Temple, 2002)
* Incapacity to discriminate colors or insufficient visual acuity that cannot be corrected
* Incapacity or unwillingness to provide informed consent
* Insufficient knowledge of French to understand and follow instructions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in subjective everyday life cognition after a 6 weeks period of gamified cognitive and physical training (program 1 vs program 2) | 6 weeks
  Subjective executive function is measured by the Working Memory Questionnaire (WMQ), a 30-item, self-administered scale (score range from 0 to 120), addressing working memory (10 items), attention (10 items) and general executive function (10 items). The higher the score, the more it reflects cognitive difficulties.
Change in speed of information processing after a 6 weeks period of gamified cognitive and physical training | 6 weeks
  Measured by the Symbol Digit Modalities Test (SDMT), scored from 0 to 110. The lower the score, the more it reflects cognitive difficulties.
Change in cognitive flexibility after a 6 weeks period of cognitive and physical training (program 1 vs program 2) | 6 weeks
  Measured by the time completion of the Color Trails Test (CTT) in CTT1 and CTT2 (i.e., Flexibility Index: (CTT2-CTT1)/CTT1). The higher the Flexibility Index, the more it reflects cognitive difficulties.
Change in visuospatial short-term memory after a 6 weeks period of cognitive and physical training (program 1 vs program 2) | 6 weeks
  Measured by the Brief Visuospatial Memory Test-Revised (BVMT-R), scored from 0 to 36. The lower the score, the more it reflects cognitive difficulties.

SECONDARY OUTCOMES:
Change in sustained attention after a 6 weeks period of gamified cognitive and physical training (program 1 vs program 2) | 6 weeks
  Measured with the Test of Variables of Attention (TOVA) using the reaction time (RT) and the false alarm rate (FA). The higher the RT and FA, the more they reflect cognitive difficulties.
Change in cognitive interference after a 6 weeks period of gamified cognitive and physical training (program 1 vs program 2) | 6 weeks
  Measured with the Denis-Kaplan Color-Word interference Stroop test using the time completion in each condition. The higher the time completion, the more it reflects cognitive difficulties.
Change in design fluency after a 6 weeks period of gamified cognitive and physical training (program 1 vs program 2) | 6 weeks
  The Five-Point Test will be used to assess design fluency using the total number of design produced. The lower the score, the more it reflects cognitive difficulties.
Change in cognitive flexibility after a 6 weeks period of gamified cognitive and physical training (program 1 vs program 2) | 6 weeks
  A subtest of a custom-made tablet-based cognitive evaluation tool will measure cognitive flexibility.
Change in visuo-spatial and verbal working memory control after a 6 weeks period of gamified cognitive and physical training (program 1 vs program 2) | 6 weeks
  Measured using the Digit and Visuo-Spatial Span Test
Change in divided attention after a 6 weeks period of gamified cognitive and physical training (program 1 vs program 2) | 6 weeks
  Measured using the Test of Attentional Performance subtest Divided Attention
Change in body composition (body fat and muscle mass) after a 6 weeks period of gamified cognitive and physical training (program 1 vs program 2) | 6 weeks
  Body composition will be measured by bioelectrical impedance measure using the percentage of body fat and muscle mass.
Change in risk of falls after a 6 weeks period of gamified cognitive and physical training (program 1 vs program 2) | 6 weeks
  Risk of falls will be assessed using the BTrackS Balance Plate (FDA registered class 1 medical device #3010668481).
Change in limits of postural stability after a 6 weeks period of gamified cognitive and physical training (program 1 vs program 2) | 6 weeks
  Limits of postural will be assessed using the BTrackS Balance Plate (FDA registered class 1 medical device #3010668481).
Change in dynamic stability after a 6 weeks period of gamified cognitive and physical training (program 1 vs program 2) | 6 weeks
  Dynamic stability will be assessed by the Four Square Step Test, which tests the participant's ability to step over objects forwards, sideways and backwards; the movements of the FSST are comparable to the ones implemented in the training program. The score is based on time taken to complete the test. The higher the score, the more it reflects balance difficulties.
Change in ability to perform a cognitive and physical dual task after a 6 weeks period of gamified cognitive and physical training (program 1 vs program 2) | 6 weeks
  In order to assess cognitive and motor dual task ability, the study participant will perform the Timed Up and Go Cognitive. The score is based on time taken to complete the test and errors or hesitations. The higher the score, the more it reflects cognitive difficulties.
Change in heart rate variability after a 6 weeks period of gamified cognitive and physical training (program 1 vs program 2) | 6 weeks
  Heart rate and heart rate variability will be recorded at rest in supine position during a 5-minute window using a medical electrocardiogramm (ECG).
Change in systolic and diastolic blood pressure after a 6 weeks period of gamified cognitive and physical training (program 1 vs program 2) | 6 weeks
  Determined by the mean of three blood pressure measurements using a sphygmomanometer and a stethoscope.
Change in anxiety after a 6 weeks period of gamified cognitive and physical training (program 1 vs program 2) | 6 weeks
  Anxiety will be assessed using the State-Trait Anxiety Inventory (STAI; 20 items) in French, scored from 20 to 80. The higher the score, the higher the level of anxiety.
Change in mood after a 6 weeks period of gamified cognitive and physical training (program 1 vs program 2) | 6 weeks
  Mood will be assessed using the Center for Epidemiologic Studies - Depression (CES-D; 20 items) in French, scored from 0 to 60. The higher the score, the higher the level of depression.
Change in everyday life activity / quality of life after a 6 weeks period of gamified cognitive and physical training | 6 weeks
  Specifically developped for patients with an HIV infection, the Medical Outcomes Study HIV Health Survey (MOS-HIV; 35 items) will be used to assess everyday life activities and health-related quality of life. The score ranges from 0 to 100. The lower the score, the poorer the quality of life.
Change in everyday life cognition after a 6 weeks period of gamified cognitive and physical training (program 1 vs program 2) | 6 weeks
  Everyday life cognition will be assessed using the Cognitive Failure Questionnaire (CFQ; 32 items). The score ranges from 0 to 128. The higher the score, the more it reflects cognitive difficulties.
Change in fatigue after a 6 weeks period of gamified cognitive and physical training (program 1 vs program 2) | 6 weeks
  Study participants will rate their degree of physical, cognitive and psychosocial fatigue on the Modified Fatigue Impact Scale (MFIS; 21 items). The score ranges from 0 to 84. The higher the score, the greater the level of fatigue.
Change in apathy after a 6 weeks period of gamified cognitive and physical training (program 1 vs program 2) | 6 weeks
  Using the self-administred Dimensional Apathy Scale (DAS; 24 items), study participants will rate their degree of apathy. The score ranges from 0 to 96. The higher the score, the greater the level of apathy.
Change in alcohol and other substance consumption after a 6 weeks period of gamified cognitive and physical training (program 1 vs program 2) | 6 weeks
  The habits in the consumption of alcohol and other substances will be evaluated with an adapted version of the Alcohol, Smoking and Substance Involvement Screening Test (ASSIST; 8 items; Khan et al, 2011).
Development of medication intake over the course of study participation. | 6 weeks
  Participants' medication intake over the course of the study will be recorded in the register of an ongoing prospective, longitudinal and multicenter study, called the Neurocognitive Assessment in the Metabolic and Aging Cohort study (NAMACO).
Development of professional occupation/employment rate over the course of study participation. | 6 weeks
  Participants' professional occupation/employment rate over the course of the study will be recorded in the register of an ongoing prospective, longitudinal and multicenter study, called the Neurocognitive Assessment in the Metabolic and Aging Cohort study (NAMACO). The employment rate will be measured in full-time equivalent, ranging from 0 to 100 %. The higher the employment rate, the better.
Development of self-reported activity profile over the course of study participation. | 6 weeks
  Participants' self-reported activity profile over the course of the study will be recorded in the register of an ongoing prospective, longitudinal and multicenter study, called the Neurocognitive Assessment in the Metabolic and Aging Cohort study (NAMACO).
Change in the theta power frequency band over the frontal brain region (Anguera et al., 2022) after a 6-week period of gamified cognitive and physical training (program 1 vs program 2) | 6 weeks
  Measured with an electroencephalogram (EEG) during the Test of Variable of Attention (TOVA).
Change in the latency of the P3b (Event-Related Potential; Anguera et al., 2013) after a 6-week period of gamified cognitive and physical training (program 1 vs program 2) | 6 weeks
  Measured with an electroencephalogram (EEG) during the TOVA.
Change in the temporal dynamic of the resting brain activity (microstates analysis; Michel and Koenig, 2018; Spring et al, 2017) after a 6-week period of gamified cognitive and physical training (program 1 vs program 2) | 6 weeks
  Measured with an electroencephalogram (EEG) during the resting state
Change in forced expiratory volume in one second (FEV1) after a 6-week period of gamified cognitive and physical training (program 1 vs program 2) | 6 weeks
  Measured by a forced exhalation in the first second of a breath into a spirometer.
Change in maximal pulmonary capacity (measured in liters) after a 6-week period of gamified cognitive and physical training (program 1 vs program 2) | 6 weeks
  Measured by a forced exhalation into a spirometer.
Change in peak oxygen capacity (VO2 peak) after a 6-week period of gamified cognitive and physical training (program 1 vs program 2) | 6 weeks
  Measure using a standardized maximal effort test with incremental exercise on a cycling ergometer with gas exchange analyses.
Change in VO2 at anaerobic threshold after a 6 weeks period of gamified cognitive and physical training (program 1 vs program 2) | 6 weeks
  VO2 at anaerobic threshold will be determined using a cyclo-ergospirometry.

OTHER OUTCOMES:
Subjective usability of the technology used in study. | 6 weeks
  Regardless of training group attribution, study participants will rate the user-friendliness of the training using the 10-item System Usability Scale scored from 0 to 40. The higher the score, the better the utility.
Subjective experience with technology used in the study | 6 weeks
  Regardless of training group attribution, study participants will rate the experience of the training using and the 4-item Perception of game training questionnaire scored from 10 to 50. The higher the score, the better the experience.
Perception of game training | 6 weeks
  Regardless of training group attribution, study participants will rate their perception of game training using the Perception of game training questionnaire (4 statements on enjoyment, challenge, frustration and motivation associated with the game, participants rate their agreement with the statement on a Likert-scale from 1 (lowest) to 7 (highest)).

CONTACTS AND LOCATIONS:
Overall Officials: Arseny A. Sokolov, Prof MD PhD, Principal Investigator — Centre Hospitalier Universitaire Vaudois (CHUV), Lausanne, Switzerland; Etienne Sallard, PhD, Study Chair — Centre Hospitalier Universitaire Vaudois (CHUV), Lausanne, Switzerland
Locations (1):
- Lausanne University Hospital (CHUV), Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Smith, A. (1982). Symbol digit modalities test (SDMT) manual (revised) Western psychological services. Los Angeles.
- [Background] Delis DC, Kramer JH, Kaplan E, Holdnack J. Reliability and validity of the Delis-Kaplan Executive Function System: an update. J Int Neuropsychol Soc. 2004 Mar;10(2):301-3. doi: 10.1017/S1355617704102191. No abstract available. PMID 15012851
- [Background] Benedict, R. H. (1997). Brief Visuospatial Memory Test-Revised (BVMT-R). Odessa, FL: Psychological Assessment Resources. In: Inc
- [Background] Vallat-Azouvi C, Pradat-Diehl P, Azouvi P. The Working Memory Questionnaire: a scale to assess everyday life problems related to deficits of working memory in brain injured patients. Neuropsychol Rehabil. 2012;22(4):634-49. doi: 10.1080/09602011.2012.681110. Epub 2012 Apr 27. PMID 22537095
- [Background] Brandt, J. (1991). The hopkins verbal learning test: Development of a new memory test with six equivalent forms. Clinical Neuropsychologist, 5(2), 125-142.
- [Background] Rieu D, Bachoud-Levi AC, Laurent A, Jurion E, Dalla Barba G. [French adaptation of the Hopkins Verbal Learning Test]. Rev Neurol (Paris). 2006 Jun;162(6-7):721-8. doi: 10.1016/s0035-3787(06)75069-x. French. PMID 16840980
- [Background] Greenberg, L., Kindschi, C., & Corman, C. (1996). TOVA clinical guide. Los Alamitos, CA: Universal Attention Disorders.
- [Background] Kollins SH, DeLoss DJ, Canadas E, Lutz J, Findling RL, Keefe RSE, Epstein JN, Cutler AJ, Faraone SV. A novel digital intervention for actively reducing severity of paediatric ADHD (STARS-ADHD): a randomised controlled trial. Lancet Digit Health. 2020 Apr;2(4):e168-e178. doi: 10.1016/S2589-7500(20)30017-0. Epub 2020 Feb 24. PMID 33334505
- [Background] Regard M, Strauss E, Knapp P. Children's production on verbal and non-verbal fluency tasks. Percept Mot Skills. 1982 Dec;55(3 Pt 1):839-44. doi: 10.2466/pms.1982.55.3.839. No abstract available. PMID 7162920
- [Background] Michel CM, Koenig T. EEG microstates as a tool for studying the temporal dynamics of whole-brain neuronal networks: A review. Neuroimage. 2018 Oct 15;180(Pt B):577-593. doi: 10.1016/j.neuroimage.2017.11.062. Epub 2017 Dec 2. PMID 29196270
- [Background] Spring JN, Tomescu MI, Barral J. A single-bout of Endurance Exercise Modulates EEG Microstates Temporal Features. Brain Topogr. 2017 Jul;30(4):461-472. doi: 10.1007/s10548-017-0570-2. Epub 2017 May 20. PMID 28528447
- [Background] Levett DZH, Jack S, Swart M, Carlisle J, Wilson J, Snowden C, Riley M, Danjoux G, Ward SA, Older P, Grocott MPW; Perioperative Exercise Testing and Training Society (POETTS). Perioperative cardiopulmonary exercise testing (CPET): consensus clinical guidelines on indications, organization, conduct, and physiological interpretation. Br J Anaesth. 2018 Mar;120(3):484-500. doi: 10.1016/j.bja.2017.10.020. Epub 2017 Nov 24. PMID 29452805
- [Background] Dite W, Temple VA. A clinical test of stepping and change of direction to identify multiple falling older adults. Arch Phys Med Rehabil. 2002 Nov;83(11):1566-71. doi: 10.1053/apmr.2002.35469. PMID 12422327
- [Background] Shumway-Cook A, Brauer S, Woollacott M. Predicting the probability for falls in community-dwelling older adults using the Timed Up & Go Test. Phys Ther. 2000 Sep;80(9):896-903. PMID 10960937
- [Background] Radloff, L. S. (1977). The CES-D Scale:A Self-Report Depression Scale for Research in the General Population. Applied Psychological Measurement, 1(3), 385-401.
- [Background] Fuhrer, R. (1989). Fuhrer, R, Rouillon F. La version française de l'échelle CES-D (Center for Epidemiologic Studies-Depression Scale). Description et traduction de l'échelle d'autoévaluation Psychiatry and Psychobiology, 4, 163-166.
- [Background] Spielberger, C. D. (1983). Manual for the State-Trait Anxiety Inventory STAI (form Y)(
- [Background] Gauthier, J., & Bouchard, S. (1993). Adaptation canadienne-française de la forme révisée du State-Trait Anxiety Inventory de Spielberger. Canadian Journal of Behavioural Science/Revue canadienne des sciences du comportement, 25(4), 559.
- [Background] Wu AW, Revicki DA, Jacobson D, Malitz FE. Evidence for reliability, validity and usefulness of the Medical Outcomes Study HIV Health Survey (MOS-HIV). Qual Life Res. 1997 Aug;6(6):481-93. doi: 10.1023/a:1018451930750. PMID 9330549
- [Background] Broadbent DE, Cooper PF, FitzGerald P, Parkes KR. The Cognitive Failures Questionnaire (CFQ) and its correlates. Br J Clin Psychol. 1982 Feb;21(1):1-16. doi: 10.1111/j.2044-8260.1982.tb01421.x. PMID 7126941
- [Background] Debouverie M, Pittion-Vouyovitch S, Louis S, Guillemin F. Validity of a French version of the fatigue impact scale in multiple sclerosis. Mult Scler. 2007 Sep;13(8):1026-32. doi: 10.1177/1352458507077942. PMID 17895294
- [Background] Fisk JD, Pontefract A, Ritvo PG, Archibald CJ, Murray TJ. The impact of fatigue on patients with multiple sclerosis. Can J Neurol Sci. 1994 Feb;21(1):9-14. PMID 8180914
- [Background] Radakovic R, Abrahams S. Developing a new apathy measurement scale: Dimensional Apathy Scale. Psychiatry Res. 2014 Nov 30;219(3):658-63. doi: 10.1016/j.psychres.2014.06.010. Epub 2014 Jun 19. PMID 24972546
- [Background] Khan R, Chatton A, Nallet A, Broers B, Thorens G, Achab-Arigo S, Poznyak V, Fleischmann A, Khazaal Y, Zullino D. Validation of the French version of the alcohol, smoking and substance involvement screening test (ASSIST). Eur Addict Res. 2011;17(4):190-7. doi: 10.1159/000326073. Epub 2011 Apr 14. PMID 21494047
- [Background] Metral M, Darling K, Locatelli I, Nadin I, Santos G, Brugger P, Kovari H, Cusini A, Gutbrod K, Tarr PE, Calmy A, Lecompte TD, Assal F, Monsch A, Kunze U, Stoeckle M, Schwind M, Schmid P, Pignatti R, Di Benedetto C, Du Pasquier R, Cavassini M; NAMACO study group; Swiss HIV Cohort Study. The Neurocognitive Assessment in the Metabolic and Aging Cohort (NAMACO) study: baseline participant profile. HIV Med. 2020 Jan;21(1):30-42. doi: 10.1111/hiv.12795. Epub 2019 Oct 7. PMID 31589807
- [Background] Brooke, J., SUS: A 'Quick and Dirty' Usability Scale. 1996.
- [Background] Boot WR, Champion M, Blakely DP, Wright T, Souders DJ, Charness N. Video games as a means to reduce age-related cognitive decline: attitudes, compliance, and effectiveness. Front Psychol. 2013 Feb 1;4:31. doi: 10.3389/fpsyg.2013.00031. eCollection 2013. PMID 23378841
- [Background] Antinori A, Arendt G, Becker JT, Brew BJ, Byrd DA, Cherner M, Clifford DB, Cinque P, Epstein LG, Goodkin K, Gisslen M, Grant I, Heaton RK, Joseph J, Marder K, Marra CM, McArthur JC, Nunn M, Price RW, Pulliam L, Robertson KR, Sacktor N, Valcour V, Wojna VE. Updated research nosology for HIV-associated neurocognitive disorders. Neurology. 2007 Oct 30;69(18):1789-99. doi: 10.1212/01.WNL.0000287431.88658.8b. Epub 2007 Oct 3. PMID 17914061
- [Background] Sheehan DV, Lecrubier Y, Sheehan KH, Amorim P, Janavs J, Weiller E, Hergueta T, Baker R, Dunbar GC. The Mini-International Neuropsychiatric Interview (M.I.N.I.): the development and validation of a structured diagnostic psychiatric interview for DSM-IV and ICD-10. J Clin Psychiatry. 1998;59 Suppl 20:22-33;quiz 34-57. PMID 9881538
- [Background] Maj M, D'Elia L, Satz P, Janssen R, Zaudig M, Uchiyama C, Starace F, Galderisi S, Chervinsky A; World Health Organization, Division of Mental Health/Global Programme on AIDS. Evaluation of two new neuropsychological tests designed to minimize cultural bias in the assessment of HIV-1 seropositive persons: a WHO study. Arch Clin Neuropsychol. 1993 Mar;8(2):123-35. PMID 14589670
- [Background] Kyle UG, Bosaeus I, De Lorenzo AD, Deurenberg P, Elia M, Gomez JM, Heitmann BL, Kent-Smith L, Melchior JC, Pirlich M, Scharfetter H, Schols AM, Pichard C; Composition of the ESPEN Working Group. Bioelectrical impedance analysis--part I: review of principles and methods. Clin Nutr. 2004 Oct;23(5):1226-43. doi: 10.1016/j.clnu.2004.06.004. PMID 15380917
- [Background] Sternberg S. High-speed scanning in human memory. Science. 1966 Aug 5;153(3736):652-4. doi: 10.1126/science.153.3736.652. PMID 5939936